CLINICAL TRIAL: NCT06570655
Title: The Study of Pharmacokinetics and Pharmacodynamics of Huperzine a Injection in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Collaborators: Zhejiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024040905
Record Dates: First submitted 2024-04-27; First posted 2024-08-26 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — huperzine A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): The same 12 subjects first received 0.2 mg single dose intravenously, then received intramuscular injection of single-dose 0.1 mg, followed by single-dose 0.2 mg, and finally single-dose 0.4 mg. A wash-out period of 7 days was applied between the doses.
  Interventions: Drug: Huperzine A injection

INTERVENTIONS:
Drug: Huperzine A injection — intramuscular
Drug: Huperzine A injection — intravenous bolus

SUMMARY:
The study used a single-center, open, sequential single-dose design. To evaluate the pharmacokinetics and dose-exposure relationship of huperzine A injection

DETAILED DESCRIPTION:
The study was divided into four modes of administration. Administration method of A: intravenous injection (non-blood collection arm), intravenous injection of 0.2mg huperzine A injection. B, C, D Administration methods: 0.1mg, 0.2mg, 0.4mg huperzine A injection was injected intramuscularly into the deltoid muscle of the upper arm (the arm on the non-blood collection side). In each cycle, after fasting for at least 10 hours, the subjects received different dosing regimens according to A sequential single dosing method, that is, each subject received dosing method A first, followed by dosing method B after the cleaning period, dosing method C after the cleaning period, and dosing method D after the cleaning period. The wash-out period between the two doses was 7 days for each subject. To evaluate the pharmacokinetics and dose-exposure relationship of huperzine A injection.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily confirms his or her willingness to participate in a particular trial and signed the written informed consent, after having been informed of all aspects of the trial that are relevant to the subject's decision to participate.They were fully aware of the adverse reactions and voluntarily signed the written informed consent.
2. The subjects were able to communicate well with the investigators and complete the trial in accordance with the protocol;
3. Gender: Chinese male or female;
4. Age: 18-45 years old (including boundary value);
5. Body mass index (BMI) 19.0-26.0 kg/m2 [BMI = weight/height 2 (kg/m2)] (including boundary values), body weight ≥50kg for men and ≥45kg for women.

Exclusion Criteria:

1. Allergic history to huperzine A or any of its components; Patients with a history of allergy to two or more drugs or foods;
2. patients who have the following clinically significant diseases at present, including but not limited to diseases of the respiratory system, circulatory system, digestive system, blood system, endocrine system, immune system, skin system, mental nervous system, ENT and other related diseases;
3. existing or suspected existing epilepsy, angina pectoris, bronchial asthma, mechanical intestinal obstruction, renal insufficiency, urinary obstruction;
4. underwent major surgical procedures within 6 months before screening or planned to undergo surgical procedures during the trial;
5. if the vital signs, physical examination, electrocardiogram and laboratory findings are clinically significant;
6. patients with a history of hepatitis B, hepatitis C, AIDS, syphilis and/or clinically significant abnormalities in one or more of the four hemodialysis tests;
7. those who had lost blood within 3 months before screening (except physiological blood loss in women) or donated blood ≥200mL or donated blood components (such as plasma, platelets, peripheral blood stem cells, etc.) within 3 months;
8. use of any drugs that alter liver enzyme activity within 30 days before screening (e.g., inductors-barbiturates, carbamazepine, phenytoin, dexamethasone, etc.; "Inhibitors - SSRI antidepressants, ciprofloxacin, diltiazem, macrolides, metronidazole, ketoconazole, verapamil.

   Rice, fluoroquinolones);
9. patients who had used any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicine) and health products within 14 days before screening, except topical drugs and eye drops;
10. vaccinated within 1 month before screening or during the planned trial period and within 1 month after the end of the trial;
11. participants who participated in a clinical trial and took a drug within 3 months before screening;
12. had a history of drug abuse within 5 years, and/or used drugs within 3 months before screening, and/or had a history of drug dependence, including herbal medicine, or screened positive for drug abuse;
13. smokers or those who did not agree to avoid using any tobacco products 48 hours before administration and during hospitalization, or who screened positive for nicotine at the first admission;
14. Regular drinkers in the preceding 6 months, defined as consuming more than 14 units of alcohol per week (1 unit =360mL of 5% beer or 45mL of 40% spirits or 150mL of 12% wine), Or did not agree to stop alcohol intake 48 hours before administration and during hospitalization, or had a positive breath alcohol test at first admission;
15. subjects who consumed excessive amounts of tea, coffee and/or caffeinated beverages (> 8 cups, 1 cup =250mL) per day before screening or disagreed with the prohibition of tea, coffee and/or caffeinated beverages 48 hours before drug administration and during hospitalization Or caffeinated foods, grapefruit (grapefruit) and/or grapefruit juice (grapefruit juice), and/or products containing poppy;
16. have a fertility plan (including sperm and egg donation plans) and/or do not agree to use an effective contraceptive method (non-drug during the trial) from the time of signing the informed consent until 3 months after the last dose of medication.

    Of;
17. difficulty in venous blood collection (unable to tolerate venipuncture, with a history of dizzy with needles and blood, poor vascular conditions, etc.);
18. subjects may not be able to complete the study for other reasons or should not be included according to the investigator's opinion.

    In addition to the above requirements, female subjects who meet the following conditions should also be excluded:
19. pregnant or lactating women or those with a positive pregnancy test;
20. who used oral contraceptives within 30 days before screening;
21. using long-acting estrogen and/or progestin injections and/or implants within 6 months before screening;
22. had unprotected sex with a partner within 14 days before screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum blood concentration of Huperzine A(Cmax) | Day1、Day8、Day15、Day22
  To measure the Cmax of Huperzine A in 4 different periods of sequential administration in 12 healthy subjects.
PK: Area under the Huperzine A blood concentration-time curve from 0min to the time of last concentration(AUC0-t) | Day1、Day8、Day15、Day22
  To measure the AUC0-t of Huperzine A in 4 different periods of sequential administration in 12 healthy subjects.
PK：Area under the Huperzine A blood concentration-time curve from 0min to the infinity time (AUC0-∞) | Day1、Day8、Day15、Day22
  To measure the AUC0-∞ of Huperzine A in 4 different periods of sequential administration in 12 healthy subjects.

SECONDARY OUTCOMES:
PD: maximum efficacy(Emax) | Day1、Day8、Day15、Day22
  Emax is defined as the maximum activities of red blood cell acetylcholinesterase and calculated as the maximum difference between erythrocyte acetylcholinesterase and baseline value. It is measured in 4 different periods of sequential administration in 12 healthy subjects.
PD: Area under the efficacy curve(AUEC) | Day1、Day8、Day15、Day22
  AUEC is defined as the area under the activity-time curve from 0min to the time of last sample collection, which is adjusted for baseline. It is measured in 4 different periods of sequential administration in 12 healthy subjects.
PD: Time to reach maximum efficacy(Tmax) | Day1、Day8、Day15、Day22
  Tmax(PD) is defined as the time to peak activity of red blood cell acetylcholinesterase. It is measured in 4 different periods of sequential administration in 12 healthy subjects.
PK: Time to peak maximum concentration of the Huperzine A(Tmax) | Day1、Day8、Day15、Day22
  Tmax(PK) is measured in 4 different periods of sequential administration in 12 healthy subjects.
PK: half life of Huperzine A(t1/2) | Day1、Day8、Day15、Day22
  t1/2 is defined as the time to eliminate half blood concentration of Huperzine A and is measured in 4 different periods of sequential administration in 12 healthy subjects.
PK: λz | Day1、Day8、Day15、Day22
  λz is defined as the blood concentration elimination rate constant of terminal phase. It is obtained by semilog linear regression with at least 3 non-zero concentration points of the end elimination phase, and the result is the inverse of the slope. It is measured in 4 different periods of sequential administration in 12 healthy subjects.
PK: Area under the curve(AUC_%Extrap) | Day1、Day8、Day15、Day22
  AUC_%Extrap is defined as the percentage of residual area which refers to the area under the Huerperzine A blood concentration-time curve. It is measured in 4 different periods of sequential administration in 12 healthy subjects.
PK: Clearance(CL) | Day1、Day8、Day15、Day22
  CL is defined as how many milliliters of Huperzine A in blood are eliminated per unit time, it is calculated by the fomula: CL=D/AUC0-∞ (D refers to the dosage of Huperzine A). It is measured in 4 different periods of sequential administration in 12 healthy subjects.
PK：Apparent volume of distribution(Vd) | Day1、Day8、Day15、Day22
  Vd is defined as the ratio of the amount of drug in the body to the concentration in the blood after the drug has reached homeostasis in the body. It is calculated by the fomula: Vd=CL/λz. It is measured in 4 different periods of sequential administration in 12 healthy subjects.
PK：Bioavailability(F) | Day1、Day8、Day15、Day22
  F is defined as the ratio of the AUC0-∞ of intramuscular administration and AUC0-∞ of intravenous administration
Urine excretion of Huperzine A.(UE) | Baseline、Day15-Day17
  UE is defined as the amout of the Huperzine A excreted in urine during the specific time. It is calculated by the fomula: UE=Cut×Vut(Cut refers to concentration of Huperzine A excreted in urine, Vut refers to the volume of urine).
Cumulative urinary excretion of Huperzine A(CUE) | Baseline、Day15-Day17
  CUE is defined as the total Huperzine A amout excreted in urine during the whole study.
Urine excretion rate(UER) | Baseline、Day15-Day17
  URE is defined as the ratio of the Huperzine A dose excreted in the urine to the dose administered during the specific time period. It is calculated by the fomula: URE=UE/D×100%(D refers to the Huperzine A administration dose)
Cumulative urinary excretion rate(CUER) | Baseline、Day15-Day17
  CURE is defined as the summary of ratio of the Huperzine A dose excreted in the urine to the dose administered during the specific time period. It is calculated by the fomula: CURE=CUE/D×100%(D refers to Huperzine A administration dose).
Faeces excretion(FE) | Baseline、Day15-Day17
  FE is defined as the amout of the Huperzine A excreted in faeces during the whole study. It is calculated by the fomula: FE=Cf×Vf(Cf refers to concentration of Huperzine A in faeces, Vf refers to the volume of faeces).
Faeces excretion rate(FER) | Baseline、Day15-Day17
  FER is defined as the ratio of the Huperzine A doses excreted in the faeces to the dose administered.It is calculated by the fomula: FER=FE/D×100%(D refers to Huperzine A administration dose).
Metabolites of Huperzine A | Day15、Day22
  To analyze the metabolites of Huperzine A by the plasma sample during the period of C and D methods administration and urine and faeces sample during the period of C method administration.(The methods of administration is explained in the detailed description)
Number of participants with adverse events (AEs) or serious adverse events (SAEs) as assessed by NCI-CTCAE v5.0. | Day1-Day28

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical trial institution of the Zhejiang Xiaoshan hospital, Hangzhou, China/Zhejiang, China

IPD SHARING:
Plan to Share IPD: No